CLINICAL TRIAL: NCT06928662
Title: Sequential Decitabine in Combination With FLAG-Ida Followed Immediately by Reduced-Intensity Conditioning (RIC) Allogeneic Hematopoietic Cell Transplantation (DEC-FLAG-Ida/RIC) for Adults With Myeloid Malignancies at High Risk of Relapse: A Phase 1/2 Study
Brief Title: Chemotherapy (Decitabine in Combination With FLAG-Ida) and Total-Body Irradiation Followed by Donor Stem Cell Transplant for the Treatment of Adults With Myeloid Malignancies at High Risk of Relapse
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG1125142; NCI-2025-01992 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); FHIRB0020797 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2025-04-08; First posted 2025-04-15 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Acute Myeloid Leukemia; Acute Undifferentiated Leukemia; Mixed Phenotype Acute Leukemia; Recurrent Acute Myeloid Leukemia; Recurrent Acute Undifferentiated Leukemia; Recurrent Chronic Myelomonocytic Leukemia; Recurrent Mixed Phenotype Acute Leukemia; Recurrent Myelodysplastic Syndrome; Refractory Acute Myeloid Leukemia; Refractory Acute Undifferentiated Leukemia; Refractory Chronic Myelomonocytic Leukemia; Refractory Mixed Phenotype Acute Leukemia; Refractory Myelodysplastic Syndrome; Secondary Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Biphenotypic, Acute; Leukemia, Myelomonocytic, Chronic; Myelodysplastic Syndromes | interventions — Decitabine; Injections; Biopsy; X-Rays; Cytarabine; Filgrastim; Granulocyte Colony-Stimulating Factor; fludarabine; Stem Cell Transplantation; Hematopoietic Stem Cell Transplantation; Idarubicin; Blood Component Removal; Whole-Body Irradiation; Specimen Handling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (decitabine, FLAG-Ida, HCT) (Experimental): DONORS: Participants undergo apheresis for collection of PBSCs on study.
  PATIENTS: Patients receive decitabine IV daily over 1 hour on days -12 to -10, -14 to -10, -16 to -10, or -19 to -10, filgrastim SC daily on days -9 to -4, idarubicin IV over 60 minutes daily on days -8 to -6, fludarabine IV over 30 minutes daily on days -8 to -4, cytarabine IV over 2 hours daily on days -8 to -4, and undergo TBI BID on day -1 or 0 OR daily on days -1 and 0 in the absence of disease progression or unacceptable toxicity. Patients then undergo HCT (receive donor PBSCs via infusion) on day 0. Patients also undergo MUGA scan or ECHO during screening, chest X-rays and bone marrow aspiration and/or biopsy during screening and as clinically indicated, and collection of blood samples throughout the study.
  Interventions: Drug: Decitabine; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Chest Radiography; Drug: Cytarabine; Procedure: Echocardiography Test; Biological: Filgrastim; Drug: Fludarabine; Procedure: Hematopoietic Cell Transplantation; Drug: Idarubicin; Procedure: Multigated Acquisition Scan; Procedure: Pheresis; Radiation: Total-Body Irradiation; Procedure: Biospecimen Collection

INTERVENTIONS:
Drug: Decitabine — Given IV
  Other Names: 5-Aza-2'-deoxycytidine; Dacogen; Decitabine for Injection; Deoxyazacytidine; Dezocitidine
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration and/or biopsies
Procedure: Bone Marrow Biopsy — Undergo bone marrow aspiration and/or biopsies
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Procedure: Chest Radiography — Undergo chest X-rays
  Other Names: Chest X-ray
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Biological: Filgrastim — Given SC
  Other Names: Filgrastim Biosimilar Filgrastim-sndz; Filgrastim Biosimilar Tbo-filgrastim; Filgrastim XM02; Filgrastim-aafi; Filgrastim-ayow; Filgrastim-sndz; G-CSF; Granix; Neupogen; Neutroval; Nivestim; Nivestym; r-metHuG-CSF; Recombinant Methionyl Human Granulocyte Colony Stimulating Factor; Releuko; rG-CSF; Tbo-filgrastim; Tevagrastim; XM02; Zarxio
Drug: Fludarabine — Given IV
  Other Names: Fluradosa
Procedure: Hematopoietic Cell Transplantation — Given via infusion
  Other Names: HCT; Hematopoietic Stem Cell Infusion; HEMATOPOIETIC STEM CELL TRANSPLANT; Hematopoietic Stem Cell Transplantation; HSCT; SCT; Stem Cell Transplant; stem cell transplantation; Stem Cell Transplantation, NOS
Drug: Idarubicin — Given IV
  Other Names: 4-Demethoxydaunomycin; 4-Demethoxydaunorubicin; 4-DMDR
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Procedure: Pheresis — Undergo apheresis
  Other Names: Apheresed; Apheresis; Blood Component Removal; Collection, Apheresis/Leukapheresis; Hemapheresis
Radiation: Total-Body Irradiation — Undergo TBI
  Other Names: SCT_TBI; TBI; Total Body Irradiation; Whole Body; Whole Body Irradiation; Whole-Body Irradiation
Procedure: Biospecimen Collection — Undergo collection of blood
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection

SUMMARY:
This phase I/II trial studies the safety, side effects, and best dose of decitabine in combination with fludarabine, cytarabine, filgrastim, and idarubicin (FLAG-Ida) and total body irradiation (TBI) followed by a donor stem cell transplant in treating adult patients with cancers of blood-forming cells of the bone marrow (myeloid malignancies) that are at high risk of coming back after treatment (relapse). Cancers eligible for this trial are acute myeloid leukemia (AML), myelodysplastic syndrome (MDS), and chronic myelomonocytic leukemia (CMML). Decitabine is in a class of medications called hypomethylation agents. It works by helping the bone marrow produce normal blood cells and by killing abnormal cells in the bone marrow. The FLAG-Ida regimen consists of the following drugs: fludarabine, cytarabine, filgrastim, and idarubicin. These are chemotherapy drugs that work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Filgrastim is in a class of medications called colony-stimulating factors. It works by helping the body make more neutrophils, a type of white blood cell. Radiation therapy uses high energy x-rays, particles, or radioactive seeds to kill cancer cells and shrink tumors. TBI is radiation therapy to the entire body. Giving chemotherapy and TBI before a donor peripheral blood stem cell (PBSC) transplant helps kill cancer cells in the body and helps make room in the patient's bone marrow for new blood-forming cells (stem cells) to grow. When the healthy stem cells from a donor are infused into a patient, they may help the patient's bone marrow make more healthy cells and platelets. Giving decitabine in combination with FLAG-Ida and TBI before donor PBSC transplant may work better than FLAG-Ida and TBI alone in treating adult patients with myeloid malignancies at high risk of relapse.

DETAILED DESCRIPTION:
OUTLINE: This is a phase I, dose-escalation study of decitabine in combination with FLAG-Ida, TBI, and HCT followed by a phase II study.

DONORS: Participants undergo apheresis for collection of PBSCs on study.

PATIENTS: Patients receive decitabine intravenously (IV) daily over 1 hour on days -12 to -10, -14 to -10, -16 to -10, or -19 to -10, filgrastim subcutaneously (SC) daily on days -9 to -4, idarubicin IV over 60 minutes daily on days -8 to -6, fludarabine IV over 30 minutes daily on days -8 to -4, cytarabine IV over 2 hours daily on days -8 to -4, and undergo TBI twice daily (BID) on day -1 or 0 OR daily on days -1 and 0 in the absence of disease progression or unacceptable toxicity. Patients then undergo HCT (receive donor PBSCs via infusion) on day 0. Patients also undergo multi-gated acquisition (MUGA) scan or echocardiography (ECHO) during screening, chest X-rays and bone marrow aspiration and/or biopsy during screening and as clinically indicated, and collection of blood samples throughout the study.

After completion of study treatment, patients are followed up at 6 months, 1 year, and 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years with an HCT-co-morbidity index (CI) ≤ 5 for patients over 60 years.
* AML (2022 World Health Organization [WHO] criteria) that is either primary refractory (as defined by failure of 2 cycles of 7+3-like chemotherapy, 1 cycle of high-dose cytarabine-based chemotherapy, or at least 2 cycles of venetoclax in combination with other therapies) or is in untreated or unsuccessfully treated first or subsequent relapse. Patients in morphologic remission (i.e. < 5% blasts in the bone marrow) but evidence of minimal residual disease (MRD) by multiparameter flow cytometry, cytogenetics/fluorescence in situ hybridization (FISH), or molecular means will be eligible for trial participation. Patients with relapsed or refractory acute leukemia of ambiguous lineage (acute undifferentiated leukemia or mixed phenotype acute leukemia) that is either primary refractory or is in untreated or unsuccessfully treated first or subsequent relapse are also eligible.
* MDS and CMML: Subjects with previously treated MDS and CMML, defined as prior treatment with at least one hypomethylating agent (hypomethylating agent [HMA]; azacitidine, decitabine and/or decitabine-cedazuridine) whose disease progressed, relapsed, or was refractory to HMA treatment as follows: 1) patients who have failed at least 4 cycles of monotherapy with azacitidine, decitabine or decitabine-cedazuridine, 2) patients who received at least 2 cycles of HMA in combination with another therapeutic agent. Subjects with MDS and CMML who failed at least 1 cycle of induction chemotherapy will be also eligible. Patients with MDS or CMML who progress to secondary AML will be eligible if they received at least 4 cycles of HMA alone or 2 cycles of HMA in combination with another therapeutic agent.
* Patients may have previously received hypomethylating agents or chemotherapy with a mitoxantrone, idarubicin- or cladribine/fludarabine-based regimen for MDS or AML. Patients who previously received up to 1 cycle of cladribine-cytarabine-filgrastim-mitoxantrone (CLAG-M) or FLAG-Ida will be eligible. Sensitivity to either CLAG-M or FLAG-Ida is not required.
* The use of hydroxyurea prior to initiation of study treatment is allowed. Patients with symptoms/signs of hyperleukocytosis, white blood cells (WBC) > 100,000/μL or with concern for other complications of high tumor burden of high tumor dynamics (e.g. disseminated intravascular coagulation) can be treated with leukapheresis or may receive up to 2 doses of cytarabine (up to 500 mg/m^2 per dose) prior to start of study treatment.
* Karnofsky score ≥ 70; Eastern Cooperative Oncology Group (ECOG) 0-1.
* Adequate cardiac function defined as absence of decompensated congestive heart failure and/or uncontrolled arrhythmia and left ventricular ejection fraction ≥ 45%.
* Bilirubin ≤ 2.5 x Institutional Upper Limit of Normal unless elevation is thought to be due to hepatic infiltration by AML, Gilbert's syndrome, or hemolysis
* Adequate pulmonary function defined as absence of oxygen (O2) requirements and either diffusion capacity of the lung for carbon monoxide (DLCO) corrected ≥ 70%mmHg or DLCO corrected 60-69%mmHg and partial pressure of oxygen (pO2) ≥ 70mmHg.
* Creatinine clearance > 60 mL/min.
* Prior autologous HCT is permissible if relapse occurred > 6 months after HCT.
* Prior TBI-containing allogeneic HCT up to 3 Gy is permissible if > 6 months after HCT.
* A human leukocyte antigen (HLA)-matched sibling/unrelated donor, mismatched unrelated donor or haploidentical donor for collection of stimulated peripheral blood stem cells must be identified and readily available.
* Ability to understand and sign a written informed consent document (or legal representative).
* SIBLING DONOR: Related to the patient and genotypically or phenotypically identical for HLA-A, B, C, DRB1 and DQB1. Phenotypic identity must be confirmed by high-resolution typing.
* MATCHED UNRELATED DONOR: Matched for HLA-A, B, C, DRB1 and DQB1 by high resolution typing; OR mismatched for a single allele without antigen mismatching at HLA-A, B, or C as defined by high resolution typing but otherwise matched for HLA-A, B, C, DRB1 and DQB1 by high resolution typing.
* MATCHED UNRELATED DONOR: Donors are excluded when preexisting immunoreactivity is identified that would jeopardize donor hematopoietic cell engraftment. The recommended procedure for patients with 10 of 10 HLA allele level (phenotypic) match is to obtain panel reactive antibody (PRA) screens to class I and class II antigens for all patients before HCT. If the PRA shows > 10% activity, then flow cytometric or B and T cell cytotoxic cross matches should be obtained. The donor should be excluded if any of the cytotoxic cross match assays are positive. For those patients with an HLA Class I allele mismatch, flow cytometric or B and T cell cytotoxic cross matches should be obtained regardless of the PRA results. A positive anti-donor cytotoxic crossmatch is an absolute donor exclusion.
* MATCHED UNRELATED DONOR: Patient and donor pairs homozygous at a mismatched allele in the graft rejection vector are considered a two-allele mismatch, i.e., the patient is A*0101 and the donor is A*0102, and this type of mismatch is not allowed.
* MISMATCHED UNRELATED DONOR: HLA-matching must be based on results of high resolution typing at HLA-A, -B, -C, -DRB1, and -DQ.
* MISMATCHED UNRELATED DONOR: Mismatch for one HLA class I antigen with or without an additional mismatch for one HLA-class I allele but matched for HLA-DRB1 and HLA-DQ.
* MISMATCHED UNRELATED DONOR: Mismatched for two HLA class I alleles but matched for HLA-DRB1 and HLA-DQ.
* MISMATCHED UNRELATED DONOR: HLA class I HLA-A, -B, -C allele matched donors allowing for any one or two DRB1 and/or DQB1 antigen/allele mismatch.
* MISMATCHED UNRELATED DONOR: If the patient is homozygous at the mismatch HLA class I locus or II locus, the donor must be heterozygous at that locus and one allele must match the patient (i.e., patient is homozygous A*01:01 and donor is heterozygous A*01:01, A*02:01). This mismatch will be considered a one-antigen mismatch for rejection only.
* HAPLOIDENTICAL DONOR: Donors must be haploidentical relatives of the patients. Donor-recipient compatibility will be tested through HLA typing at high resolution for the HLA loci (-A, -B, -C, -DRB1, -DQB1). Donor and recipient should share at least 5/10 HLA loci.
* HAPLOIDENTICAL DONOR: Age ≥ 18 years.
* HAPLOIDENTICAL DONOR: Weight ≥ 40 kg.
* HAPLOIDENTICAL DONOR: Donor must meet the selection criteria as defined by the Foundation of the Accreditation of Cell Therapy (FACT) and will be screened per the American Association of Blood Banks (AABB) guidelines.
* DONOR: In case of more available donors, selection criteria should include, in this order:

  * For cytomegalovirus (CMV) seronegative recipients, a CMV seronegative donor
  * Red Blood Cell compatibility

    * Red blood cell (RBC) cross match compatible
    * Minor ABO incompatibility
    * Major ABO incompatibility
* DONOR: Donors will undergo diagnostic evaluation (clinical, laboratory test and imaging) as indicated per institutional guidelines.

Exclusion Criteria:

* Active central nervous system (CNS) disease.
* Concomitant illness associated with a likely survival of < 1 year.
* Active systemic fungal, bacterial, viral, or other infection, unless disease is under treatment with antimicrobials and/or controlled or stable. Patients with fever thought to be likely secondary to myeloid malignancy are eligible.
* Known hypersensitivity or contraindication to any study drug used in this trial.
* Pregnancy or lactation.
* Concurrent treatment with any other approved or investigational anti-leukemia agent.
* HAPLOIDENTICAL DONOR: Since detection of anti-donor-specific antibodies (anti-DSA) is associated with higher graft rejection rate, patients will be screened for anti-DSA pre-transplant. Patient with DSA mean fluorescent intensity (MFI) < 5000 after desensitization treatment, will be considered eligible to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-09-23 (Actual); Primary Completion 2028-03-09 (Estimated); Study Completion 2028-11-29 (Estimated)

PRIMARY OUTCOMES:
Non-relapse mortality (Phase 1) | At day 100
  Will evaluate whether intensification of fludarabine, cytarabine, filgrastim, and idarubicin/reduced intensity conditioning with the potential sequential addition of 4 escalating doses of decitabine prior to allografting with 4 Gy total-body irradiation would be feasible with an acceptable rate of toxicity and non-relapse mortality within the first 100 days following allograft, where day -100 non-relapse mortality is meant to encompass various measures of "toxicity".
Disease-free survival (Phase 2) | At 1 year

SECONDARY OUTCOMES:
Rate of stem cell engraftment (Phase 1) | Up to day 80
  Will use exploratory, descriptive, and observational methods to 1) estimate the rates of stem cell engraftment.
Rate of donor chimerism (Phase 1) | Up to day 80
  Will use exploratory, descriptive, and observational methods to estimate donor chimerism.
Rates of grades II-IV acute graft-versus-host disease (GVHD) (Phase 1) | Up to 2 years
  Will use exploratory, descriptive, and observational methods to estimate the rates of grades II-IV acute GVHD requiring systemic immunosuppressive treatment.
Rates of grades II-IV chronic GVHD (Phase 1) | Up to 2 years
  Will use exploratory, descriptive, and observational methods to estimate the rates of grades II-IV chronic GVHD requiring systemic immunosuppressive treatment.
Disease response (Phase 1) | Up to 2 years
  Will use exploratory, descriptive, and observational methods to estimate disease response.
Duration of remission (Phase 1) | Up to 2 years
  Will use exploratory, descriptive, and observational methods to estimate duration of remission.

CONTACTS AND LOCATIONS:
Overall Officials: Naveed Ali, MD, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No